CLINICAL TRIAL: NCT06410261
Title: Randomized Pilot Study Evaluating the Effect of a 6-Month Exercise Rehabilitation Program on Physical and Cognitive Function in Persons With MS Who Use Wheelchairs as a Primary Mobility Device
Brief Title: Exercise Rehabilitation Program in MS Who Use Wheelchairs as a Primary Mobility Device
Acronym: MSGH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Enrico Benedetti, Department Head, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY2024-0273
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis
Keywords: Exercise; Rehabilitation; Physical function; Cognition
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise rehabilitation program (Experimental): • Participants will take part in a personalized, one-hour, one-on-one muscle therapy session, two days a week, for 6 months.
  Interventions: Behavioral: Exercise rehabilitation program
- Control (No Intervention): • Participants will complete the study measures on three separate occasions and will have the option to complete the exercise rehabilitation intervention once the study reaches completion.

INTERVENTIONS:
Behavioral: Exercise rehabilitation program — * The sessions will consist of a customized low-impact, resistance-base rehabilitation regime to increase muscle strength and functionality by focusing on isolating each targeted muscle, without increasing the participant's fatigue or pain level.
  * The goal of phase one will be to start muscle activation without increasing fatigue or pain. Low intensity, single set of 30-35 repetitions for each of the targeted muscles will be performed by the participants, followed by stretching; the goal of phase two will be to progressively develop muscle strength, without increasing pain or fatigue. A single set of 20-25 repetitions for each muscle will be prescribed, followed by stretching; during phase three, the emphasis will be on further development of muscle strength, function, and endurance.
  Other Names: GH Method
  Arms: Exercise rehabilitation program

SUMMARY:
Approximately 50% of people with multiple sclerosis (MS) use a wheelchair within 30 years of the initial diagnosis. Wheelchair use in MS is often associated with fatigue as a consequence of muscle weakness. Indeed, fatigue, a prevalent consequence of MS, often becomes debilitating and exhausts energetic resources when carrying-out tasks of daily life and/or interacting with the community, as these require ambulatory mobility. This experience of excessive fatigue has its roots in muscle weakness and results in reliance on a wheelchair for mobility, and the dependency on a wheelchair may further reduce muscular strength, particularly of the lower extremities. We propose that wheelchair users with MS can increase muscular strength through a personalized exercise rehabilitation, and this in turn will improve ambulatory performance and possibly reduce fatigue. To date, no research has examined the effects of this specific exercise rehabilitation program (GH method) on physical function and other disease-related outcomes in persons with MS who use wheelchairs as a primary mobility device.

DETAILED DESCRIPTION:
To date, there is a dearth of clinical trials examining exercise programs targeting wheelchair users with MS, but exercise programs are ideally suited for targeting the underlying causes of wheelchair use in this population, namely reduced lower extremity strength that manifests as excessive fatigue when undertaking tasks of daily life and/or interacting with the community. We propose examining a novel and highly relevant exercise rehabilitation program (GH method) on physical function and other disease-related outcomes in persons with MS who use wheelchairs as a primary mobility device.

There are no relevant preliminary data in wheelchair users with MS, but the GH method has been successfully applied in other chronic, disabling diseases such as chronic kidney disease (CKD). The data from our previous and ongoing application of GH in CKD has supported improvements in a range of outcomes from physical frailty through quality of life.

This proposed research will test the effects of a 6-month exercise rehabilitation program on physical function, self-reported health-related outcomes, and cognitive function in persons with MS who use wheelchairs as a primary mobility device in the community, but who are still ambulatory. These findings may guide researchers, clinicians, and exercise specialists in the advancement of future interventions for improving the lives of persons from this segment of the population with MS.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS
* age above 18 years
* no relapse within last 30 days
* use of wheelchair for mobility in the community
* ability to walk at least 50 feet (or 65 steps) using an assistive device
* low risk for contraindications of physical activity indicated by no more than a single "yes"
* response on the Physical Activity Readiness Questionnaire (PAR-Q)
* willingness to complete the assessments and undergo randomization

Exclusion Criteria:

* no diagnosis of MS
* less than 18 years of age
* not relapse-free within the last 30 days
* no use of wheelchair as primary mobility device
* no ability to walk for at least 50 feet (or 65 steps)
* high risk for contraindications based on more than a single "yes" response on the PAR-Q
* not willing to complete the testing procedures and undergo randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical Function | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Short Physical Performance Battery (SPPB); the performance scores range between 0 (min) and 12 (max) points, higher scores reflect better physical function
Walking Speed | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Timed 25-foot Walking Test (T25FW); the score is the average speed (25 feet divided by time, ft/s) for completing two trials. The minimum and maximum scores (time) depend on individuals' performance. A faster speed represents better ambulatory performance
Lower-Extremity Function | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  30-Second Sit to Stand Test (30STS). The score is the number of complete repetitions of sit-to-stand movements performed during 30 seconds; the minimum value is 0 repetitions, and the maximum value depends on individuals' performance. Higher scores reflect better lower extremity function
Walking Endurance | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Six-Minute Walk Test (6MW); the score is the total walking distance (in meters) during the 6 minutes. The minimum value is 0 meter, and the maximum value depends on individuals' performance. A longer distance (higher scores) indicates better walking endurance

SECONDARY OUTCOMES:
Cognitive Function | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Symbol Digits Modalities Test (SDMT); the total test scores range between 0 (min) and 110 (max), higher scores indicate better cognitive function
Cognitive Function | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  California Verbal Learning Test - Second Edition (CVLT-II); the total test scores range between 0 (min) and 80 (max), higher scores indicate better cognitive function
Fatigue Severity | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Fatigue Severity Scale (FSS); scores range between 1 (min) and 7 (max), higher scores reflect greater fatigue severity
Fatigue Impact | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Modified Fatigue Impact Scale (MFIS); scores range between 0 (min) and 84 (max), higher scores reflect a greater impact of fatigue on daily life
Depressive Symptoms | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms
Anxiety | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Hospital Anxiety and Depression Scale (HADS); scores range between 0 (min) and 21 (max), higher scores reflect greater frequency of anxiety and depressive symptoms
Health-Related Quality of Life | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Multiple Sclerosis Impact Scale (MSIS-29); scores range between 0 (min) and 100 (max), higher scores indicate greater impact of disease on daily function (i.e. worse outcomes)
Exercise Behavior | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  Godin Leisure-Time Exercise Questionnaire (GLTEQ); scores range between 0 (min) and 119 (max), higher scores indicate greater engagement in exercise behavior
Usual Pattern of Mobility in Various Life-Space Levels | Changes in physical function scores from Baseline (pre-intervention), after 3 months (mid-intervention), and after 6 months (post-intervention)
  The University of Alabama at Birmingham Study of Aging Life-Space Assessment (UAB-LSA); scores range between 0 (min) and 120 (max), higher scores indicate better mobility in various life-space levels

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Benedetti, MD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No